CLINICAL TRIAL: NCT00471263
Title: The Effects of Casigold and Casimax on Blood Pressure in Subjects With Highnormal Blood Pressure or Mild Hypertension
Brief Title: The Effects of Milk Proteins on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: DSM Food Specialties (Industry)
Responsible Party: Dr. J. Kloek, DSM Food Specialties
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P7365
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Casigold
Drug: Casimax
Drug: Placebo

SUMMARY:
The primary purpose of the study is to demonstrate a blood pressure lowering effect of CasiGold and CasiMax in subjects with high-normal blood pressure or mild hypertension. The secondary purpose is to collect human safety data after treatment with CasiGold and CasiMax, to gain insight into potential mechanisms by measurement of renin and angiotensin I and II, and to evaluate the genetic determinants of the individual BP lowering response by measurement of specific genetic polymorphisms.

DETAILED DESCRIPTION:
Rationale: Hypertension is the major controllable risk factor associated with cardiovascular disease. The risk of developing CVD is directly related to blood pressure (BP) level. Tripeptides IPP and VPP obtained from milk proteins were shown to have potential blood lowering effects. The renin-angiotensin system is one of the major pathways of BP regulation, and ACE inhibition is an important target for BP control. CasiGold and CasiMax are hydrolysed casein preparations consisting of relatively high concentrations tripeptides which have ACE inhibitory properties in vitro and which may have beneficial effects on blood pressure.

Study population: 84 female and male Caucasians with a high-normal blood pressure or mild hypertension, aged 30 - 70 years at Day 01 of the study and with a BMI 18 - 32 kg/m2, will participate in the study.

Intervention: All subjects receive all treatments, but in a different order. One of the treatments consists of daily consumption of two capsules Casigold containing IPP during a period of 4 weeks. One of the treatments consists of daily consumption of two capsules Casimax containing a mixture of tripeptides during a period of 4 weeks. And one of the treatments consists of daily consumption of two capsules placebo during a period of 4 weeks. One capsule will be taken upon completion of breakfast and one capsule will be taken upon completion of dinner.

Main study parameters: The main study parameter is the blood pressure after 4 weeks of each treatment. Blood pressure will be measured at the study site on the two last days of each treatment period. Other study parameters include evaluation of safety at the end of each treatment period, and determination of genetic polymorphisms. Analysis of renin and angiotensin I and II will only be done in case a change in BP is found.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male Caucasians
* Age between 30 and 70 years at Day 01 of the study
* Body Mass Index (BMI) 18 - 32 kg/m2
* Blood pressure: SBP 120-139 mmHg/DBP 80-89 mmHg (pre-hypertension) or SBP 140-159/DBP 90-99 mmHg (stage 1 hypertension)
* Voluntary participation
* Having given their written informed consent
* Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
* Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Having a history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease or systolic blood pressure ≥ 160 mm Hg after repeated measurements
* Any concomitant medication, with the exception of paracetamol, that may influence the outcome of the study
* Intolerance or allergy to milk products
* Not willing to give up consumption of >1 fermented dairy product per day
* Alcohol consumption > 28 units/week for males or > 21 units/week for females women)
* Smoking
* Reported unexplained weight loss or weight gain of > 2 kg in the month prior to pre-study screening or during the study
* Reported slimming or medically prescribed diet
* Reported vegan, vegetarian or macrobiotic life-style
* Participation in night shift work
* Pregnant or lactating or wishing to became pregnant in the period of the study
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding a subject's health to and from a subject's general practitioner.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-05-07 (Actual); Primary Completion 2007-12-18 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 4 weeks

SECONDARY OUTCOMES:
Safety data in blood and urine | 4 weeks
Genetic determinants of the individual BP lowering response by measurement of specific genetic polymorphisms. | once during the study
Potential mechanisms by measurement of renin and angiotensin I and II (only be done in case a change in BP is found). | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Esther Boelsma, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Netherlands

REFERENCES:
- [Derived] Boelsma E, Kloek J. IPP-rich milk protein hydrolysate lowers blood pressure in subjects with stage 1 hypertension, a randomized controlled trial. Nutr J. 2010 Nov 8;9:52. doi: 10.1186/1475-2891-9-52. PMID 21059213